CLINICAL TRIAL: NCT01148108
Title: Phase 2 Study of Canfosfamide HCl for Injection (Telcyta®, TLK286)in Refractory or Relapsed Mantle Cell Lymphoma (MCL), Diffuse Large B Cell Lymphoma (DLBCL) and Multiple Myeloma (MM)
Brief Title: Study of Canfosfamide in Refractory or Relapsed Mantle Cell, Diffuse Large B Cell Lymphoma and Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Telik (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TLK286.2030
Record Dates: First submitted 2010-06-17; First posted 2010-06-22 (Estimated); Last update posted 2013-03-15 (Estimated); Status verified 2013-03

CONDITIONS: Mantle Cell Lymphoma; B Cell Lymphoma; Multiple Myeloma
Keywords: NHL; Non-Hodgkins Lymphoma; Lymphoma; Mantle Cell; Diffuse Large B Cell; Multiple Myeloma; Telcyta; canfosfamide; TLK286; Prodrug; Enzyme activated drug; Glutathione Transferase P1-1 activated drug; GSTp1-1 activated drug; Glutathione Transferase activated drug; Glutathione; Glutathione analong
MeSH Terms: conditions — Lymphoma, Mantle-Cell; Lymphoma, B-Cell; Multiple Myeloma; Lymphoma, Non-Hodgkin; Lymphoma | interventions — TER 286; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Mantle Cell Lymphoma (Experimental): Patients with relapsed or refractory mantle cell lymphoma
  Interventions: Drug: Canfosfamide HCl for injection
- Diffuse Large B Cell Lymphoma (Experimental): Patients with relapsed or refractory diffuse large B cell lymphoma
  Interventions: Drug: Canfosfamide HCl for injection
- Multiple Myeloma (Experimental): Patients with relapsed or refractory multiple myeloma
  Interventions: Drug: Canfosfamide HCl for injection

INTERVENTIONS:
Drug: Canfosfamide HCl for injection — 30 min. intravenous infusion of canfosfamide HCl (1000 mg/m2) every 2 weeks
  Other Names: Telcyta; TLK286

SUMMARY:
This is a Phase 2 study to determine the efficacy and safety of canfosfamide treatment in relapsed or refractory mantle cell lymphoma, diffuse large B cell lymphoma and multiple myeloma. The study will be conducted in two stages with 5-6 patients in each indication in Stage 1 and if responses are observed an additional 10 patients in Stage 2 in each group.

ELIGIBILITY:
Inclusion Criteria:

* relapsed or refractory disease
* histologically or cytologically confirmed disease
* characteristic immunophenotypic profiles
* measurable disease (for lymphoma patients)
* ECOG performance status of 0-2
* adequate liver and kidney function
* adequate bone marrow reserves
* ineligible or unwilling to undergo autologous stem cell transplantation

Exclusion Criteria:

* failure to recover from any major surgery within 4 weeks of study entry
* pregnant or lactating women
* women of child-bearing potential not using reliable and appropriate contraception
* routine prophylactic use of G-CSF required within 2 weeks of study entry
* Grade 3 or higher peripheral neuropathy
* history of hepatitis B virus or HIV
* central nervous system or meningeal involvement by lymphoma or multiple myeloma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2010-06; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate | At 6 weeks of treatment
  Disease will be assessed every 6 weeks using International Working Group Response Criteria for Non-Hodgkins Lymphoma in the mantle cell and diffuse large B cell lymphoma patients and the International Myeloma Working Group Response Criteria for multiple myeloma patients. Patients will continue to be treated and disease assessed until disease progression or unacceptable toxicity.
Objective Response Rate | At 12 weeks of treatment
  Disease will be assessed every 6 weeks using International Working Group Response Criteria for Non-Hodgkins Lymphoma in the mantle cell and diffuse large B cell lymphoma patients and the International Myeloma Working Group Response Criteria for multiple myeloma patients. Patients will continue to be treated and disease assessed until disease progression or unacceptable toxicity.
Objective Response Rate | At 18 weeks of treatment
  Disease will be assessed every 6 weeks using International Working Group Response Criteria for Non-Hodgkins Lymphoma in the mantle cell and diffuse large B cell lymphoma patients and the International Myeloma Working Group Response Criteria for multiple myeloma patients. Patients will continue to be treated and disease assessed until disease progression or unacceptable toxicity.
Objective Response Rate | At 24 weeks of treatment
  Disease will be assessed every 6 weeks using International Working Group Response Criteria for Non-Hodgkins Lymphoma in the mantle cell and diffuse large B cell lymphoma patients and the International Myeloma Working Group Response Criteria for multiple myeloma patients. Patients will continue to be treated and disease assessed until disease progression or unacceptable toxicity.

SECONDARY OUTCOMES:
Duration of Response | At 6, 12, 18 & 24 weeks of treatment
  Duration of response will be determined after disease progression is documented in patients who have an objective response.
Safety Assessments | At 3, 6, 9, & 12 weeks of treatment
  Toxicity will be assessed throughout study using the National Cancer Institute Common Terminology Criteria for Adverse Events Version 3.0.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Bertino, MD, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (1):
- Cancer Institute of New Jersey, New Brunswick, New Jersey, United States